CLINICAL TRIAL: NCT00875485
Title: An Open Multicentre, Multicountry Study to Evaluate Long-term Antibody Persistence and Immune Memory Between Years 11 and 15 After the Primary Study HAB-084 in Which Healthy Adolescents Were Vaccinated With Twinrix™ Adult Following a Two-dose Schedule or Twinrix™ Junior Following a Three-dose Schedule.
Brief Title: Evaluation of Antibody Persistence & Immune Memory in Subjects Vaccinated During Adolescence With Twinrix™
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 110699; 110700 (Other: GSK); 110701 (Other: GSK); 110702 (Other: GSK); 110703 (Other: GSK); 110704 (Other: GSK)
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Results first posted 2010-07-05 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-07

CONDITIONS: Hepatitis B; Hepatitis A
Keywords: Monovalent Hepatitis A; hepatitis B vaccine; Belgium and Czech Republic
MeSH Terms: conditions — Hepatitis B; Hepatitis A | interventions — Blood Specimen Collection

ARMS (2):
- Twinrix Adult Group (Experimental): Subjects received 2 doses of Twinrix™ Adult intramuscularly according to a 0, 6 month schedule in the primary study
  Interventions: Procedure: Blood sampling; Biological: Additional challenge dose
- Twinrix Junior Group (Experimental): Subjects received 3 doses of Twinrix™ Junior (= half dose Twinrix™ Adult) intramuscularly according to a 0, 1, 6 month schedule in the primary study
  Interventions: Procedure: Blood sampling; Biological: Additional challenge dose

INTERVENTIONS:
Procedure: Blood sampling — Blood sampling at Years 11, 12, 13, 14, 15 and at the time of challenge dose administration and one month after challenge dose administration.
Biological: Additional challenge dose — If a subject became seronegative for anti-HAV antibodies (< 15 mIU/mL) or if anti-HBs antibody concentrations decreased below 10 mIU/mL during the long-term follow-up, immune memory against the antigen was evaluated by administering a challenge dose of the appropriate antigen (vaccine) 6 to 12 months after the Year 15 follow-up time-point.

SUMMARY:
This study will evaluate the immune response against Hepatitis-A (HAV) and Hepatitis B surface (HBs) antigen in healthy subjects aged 12 to 15 years (at the time of primary vaccination), who received vaccination course with GSK Biologicals' Twinrix Adult and Twinrix Junior vaccine, approximately 10 years ago in the primary study. The subjects will be invited for blood sampling at 11, 12, 13, 14 and 15 years after primary vaccination to evaluate the persistence of immune response. For subjects detected with decreased immunity, the presence of immune memory against hepatitis A & B antigens will be investigated by the administration of a challenge dose of the appropriate vaccine 6 to 12 months after the Year 15 follow-up time-point.

No new subjects will be recruited during this booster phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female who received the complete primary vaccination course according to his/her group allocation in the primary study
* Written informed consent obtained from the subject.

All subjects must satisfy the following criteria at entry into the challenge dose phase:

* A male or female who received the complete primary vaccination course according to his/her group allocation in the primary study.
* Subjects who participated in the long-term follow-up phase of the primary study and for whom the antibody concentrations were below specified value for anti-HAV antibodies and/ or for anti-HBs antibodies at the last available follow-up time-points.
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* Written informed consent obtained from the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the challenge dose phase of this study.
* If the subject is female, she must be of non-childbearing potential, i.e. either surgically sterilized; or, if of childbearing potential, she must be abstinent or have used adequate contraceptive precautions for 30 days prior to vaccination, have a negative pregnancy test and must agree to continue such precautions for two months after the vaccination.

Exclusion Criteria:

The following criteria should be checked at each follow-up visit. If any apply at study entry, the subject must not be included at that long-term follow-up visit.

* Use of any investigational or non-registered product (drug or vaccine) since the last blood sampling visit.
* Administration of a hepatitis A, hepatitis B or hepatitis combination vaccine since the primary vaccination course of the primary study.
* History of hepatitis A or hepatitis B infection.
* Administration of hepatitis A or hepatitis B immunoglobulins and/or any blood products within 3 months prior to blood sampling.

The following criteria should be checked before the challenge dose phase. If any apply, the subject must not be included in the challenge dose phase:

* Use of any investigational or non-registered product (drug or vaccine) within 30 days before the administration of the challenge dose or planned use during the study period outside the context of the study.
* Administration of a hepatitis A, hepatitis B or hepatitis combination vaccine between the primary vaccination course of the primary study and the challenge dose visit.
* History of hepatitis A or hepatitis B infection.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the challenge dose.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* Acute disease at the time of.
* Administration of immunoglobulins and/or any blood products within the three months preceding the administration of the challenge dose or planned administration before the final blood sampling point (one month after the challenge dose).
* Pregnant or lactating female.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 210 (Actual)
Dates: Start 2009-05-01; Primary Completion 2014-07-01 (Actual); Study Completion 2014-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Brussels, Belgium
- GSK Investigational Site, Hradec Králové, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Agrawal A, Kolhapure S, Andani A, Ota MOC, Badur S, Karkada N, Mitra M. Long-Term Persistence of Antibody Response with Two Doses of Inactivated Hepatitis A Vaccine in Children. Infect Dis Ther. 2020 Dec;9(4):785-796. doi: 10.1007/s40121-020-00311-8. Epub 2020 Jul 24. PMID 32710245
- [Derived] Beran J, Van Der Meeren O, Leyssen M, D'silva P. Immunity to hepatitis A and B persists for at least 15 years after immunisation of adolescents with a combined hepatitis A and B vaccine. Vaccine. 2016 May 23;34(24):2686-91. doi: 10.1016/j.vaccine.2016.04.033. Epub 2016 Apr 20. PMID 27105563
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 110699 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110699 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110699 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110699 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110699 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this study, a total of 210 subjects were enrolled who participated at Year 11 (Y11) and Y12. There were a total of 8 additional subjects at Y13 and Y14 who came back from the primary study but did not participate in Y11 and Y12 as allowed by the protocol. One subject from the 210 subjects who participated in Y11 and Y12 did not return at Y15.
Period: Year 11
Arm/Group | Twinrix Adult Group | Twinrix Junior Group
Started | 99 | 111
Completed | 99 | 111
Not Completed | 0 | 0
Period: Year 12
Arm/Group | Twinrix Adult Group | Twinrix Junior Group
Started | 101 | 109
Completed | 101 | 109
Not Completed | 0 | 0
Period: Year 13
Arm/Group | Twinrix Adult Group | Twinrix Junior Group
Started | 102 | 113
Completed | 102 | 113
Not Completed | 0 | 0
Period: Year 14
Arm/Group | Twinrix Adult Group | Twinrix Junior Group
Started | 100 | 113
Completed | 100 | 113
Not Completed | 0 | 0
Period: Year 15
Arm/Group | Twinrix Adult Group | Twinrix Junior Group
Started | 98 | 111
Completed | 98 | 111
Not Completed | 0 | 0
Period: Challenge Dose Epoch
Arm/Group | Twinrix Adult Group | Twinrix Junior Group
Started | 8 | 11
Completed | 7 | 11
Not Completed | 1 | 0
Not completed — Pregnancy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Twinrix Adult Group | Twinrix Junior Group | Total
Number analyzed (Participants) | 102 | 113 | 215
Age, Continuous [Mean (Standard Deviation); unit: years] — The baseline measure data here corresponds to Year 11. Population: The analysis Population includes all subjects that returned for the Year 11 follow up time point.
  years
    number analyzed (Participants) | 99 | 111 | 210
    (all) | 24.5 (1.06) | 24.5 (1.05) | 24.5 (1.05)
Age, Continuous [Mean (Standard Deviation); unit: Years] — The baseline measure data here corresponds to Year 12 Population: The analysis Population includes all subjects that returned for the Year 12 follow up time point.
  Years
    number analyzed (Participants) | 101 | 109 | 210
    (all) | 25.4 (1.06) | 25.4 (1.04) | 25.40 (1.05)
Age, Continuous [Mean (Standard Deviation); unit: Years] — The baseline measure data here corresponds to Year 13 Population: The analysis Population includes all subjects that returned for the Year 13 follow up time point.
  Years | 26.40 (1.07) | 26.4 (1.06) | 26.40 (1.06)
Age, Continuous [Mean (Standard Deviation); unit: Years] — The baseline measure data here corresponds to Year 14 Population: The analysis Population includes all subjects that returned for the Year 14 follow up time point.
  Years
    number analyzed (Participants) | 100 | 113 | 213
    (all) | 27.40 (1.11) | 27.40 (1.05) | 27.40 (1.08)
Age, Continuous [Mean (Standard Deviation); unit: Years] — The baseline measure data here corresponds to Year 15 Population: The analysis Population includes all subjects that returned for the Year 15 follow up time point.
  Years
    number analyzed (Participants) | 98 | 111 | 209
    (all) | 28.4 (1.15) | 28.3 (1.09) | 28.3 (1.12)
Age, Continuous [Mean (Standard Deviation); unit: Years] — The baseline measure data here corresponds to the challenge dose epoch Population: The analysis Population includes all subjects that were administrated a challenge dose.
  Years
    number analyzed (Participants) | 8 | 11 | 19
    (all) | 29.4 (1.2) | 29.4 (1.3) | 29.4 (1.22)
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to Year 11. Population: The analysis Population includes all subjects that returned for the Year 11 follow up time point.
  Participants
    number analyzed (Participants) | 99 | 111 | 210
    Female | 49 | 52 | 101
    Male | 50 | 59 | 109
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to Year 12 Population: The analysis Population includes all subjects that returned for the Year 12 follow up time point.
  Participants
    number analyzed (Participants) | 101 | 109 | 210
    Female | 50 | 50 | 100
    Male | 51 | 59 | 110
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to Year 13 Population: The analysis Population includes all subjects that returned for the Year 13 follow up time point.
  Participants
    Female | 50 | 53 | 103
    Male | 52 | 60 | 112
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to Year 14 Population: The analysis Population includes all subjects that returned for the Year 14 follow up time point.
  Participants
    number analyzed (Participants) | 100 | 113 | 213
    Female | 49 | 53 | 102
    Male | 51 | 60 | 111
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to Year 15 Population: The analysis Population includes all subjects that returned for the Year 15 follow up time point.
  Participants
    number analyzed (Participants) | 98 | 111 | 209
    Female | 47 | 52 | 99
    Male | 51 | 59 | 110
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to the challenge dose epoch Population: The analysis Population includes all subjects that were administrated a challenge dose.
  Participants
    number analyzed (Participants) | 8 | 11 | 19
    Female | 4 | 7 | 11
    Male | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Anti-HAV Antibody Concentrations
Description: Antibody concentrations are expressed as Geometric Mean Concentrations (GMCs) in mIU/mL. The analysis was performed on anti-HAV seropositive subjects. Seropositive subjects are subjects with anti-HAV antibody concentrations >= 15 mIU/mL.
Time Frame: At Year 11, 12, 13, 14 and 15 after the first vaccine dose of two-dose or three-dose primary vaccination in study HAB-084
Population: Analysis was performed on subjects from the Long Term According-to-Protocol (LT ATP) cohort for immunogenicity on anti-HAV seropositive subjects with available data at the specified time-points.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Twinrix Adult Group | Twinrix Junior Group
Number analyzed (Participants) | 78 | 92
mIU/mL
  Year 11 (N= 78; 92) | 360.5 [292.0 to 445.1] | 257.2 [215.1 to 307.5]
  Year 12 (N= 75; 90) | 450.8 [359.6 to 565.1] | 335.6 [279.0 to 403.6]
  Year 13 (N= 77; 92) | 401.5 [328.2 to 491.1] | 293.6 [244.2 to 352.9]
  Year 14 (N= 75; 91) | 388.0 [309.2 to 487.0] | 291.4 [240.6 to 352.9]
  Year 15 (N= 74; 88) | 387.5 [306.6 to 489.8] | 299.4 [247.6 to 362.0]

2. Primary Outcome: Number of Subjects With Anti-Hepatitis B Surface Antigen (HBs) Antibody Concentrations Equal to or Above the Cut-Off Values
Description: Anti-HBs antibody cut-off values assessed were >= 6.2 mIU/mL and >= 10 mIU/mL. Note: A decrease in the specificity of the anti-HB ELISA assay had been observed in some studies for low levels of antibody (10-100 mIU/mL). The table shows updated results following complete retesting and reanalysis for years 11 to 13. Results of year 14 and year 15 were only analysed by ChemiLuminescence ImmunoAssay (CLIA).
Time Frame: At Year 11, 12, 13, 14 and 15 after the first vaccine dose of the two-dose or three-dose primary vaccination in study HAB-084
Population: Analysis was performed on subjects from the Long Term According-to-Protocol (LT ATP) cohort for immunogenicity on subjects with available data at the specified time-points
Measure: Number; unit: Subjects
Arm/Group | Twinrix Adult Group | Twinrix Junior Group
Number analyzed (Participants) | 78 | 92
Subjects
  Year 11 [6.2 mIU/mL] (N = 78;91) | 68 | 79
  Year 12 [6.2 mIU/mL] (N = 75;90) | 64 | 80
  Year 13 [6.2 mIU/mL] (N = 77;92) | 65 | 83
  Year 14 [6.2 mIU/mL] (N= 75;91) | 66 | 80
  Year 15 [6.2 mIU/mL] (N= 74;88) | 62 | 79
  Year 11 [10 mIU/mL] (N = 78;91) | 64 | 75
  Year 12 [10 mIU/mL] (N = 75;90) | 62 | 76
  Year 13 [10 mIU/mL] (N = 77;92) | 62 | 77
  Year 14 [10 mIU/mL] (N= 75;91) | 62 | 73
  Year 15 [10 mIU/mL] (N= 74;88) | 60 | 72

3. Primary Outcome: Anti-HBs Antibody Concentrations
Description: Antibodys concentrations are expressed as Geometric Mean concentrations (GMCs) in mIU/mL. The analysis was performed on anti-HBs seropositive subjects. Seropositive subjects are subjects with anti-HBs antibody concentrations >= 6.2 mIU/mL.
  Note: A decrease in the specificity of the anti-HB ELISA assay had been observed in some studies for low levels of antibody (10-100 mIU/mL). The table shows updated results following complete retesting and reanalysis for years 11 to 13. Results of year 14 and year 15 were only analysed by CLIA.
Time Frame: At Year 11, 12, 13, 14 and 15 after the first vaccine dose of a two-dose or a three-dose primary vaccination in study HAB-084.
Population: Analysis was performes on subjects from the Long Term According-to-Protocol (LT ATP) cohort forimmunogenicity on anti-HBs seropositive subjects with available data at the specified time-points.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Twinrix Adult Group | Twinrix Junior Group
Number analyzed (Participants) | 78 | 92
mIU/mL
  Year 11 (N = 78;91) | 88.0 [63.2 to 122.5] | 75.2 [55.6 to 101.8]
  Year 12 (N = 75;90) | 93.3 [66.2 to 131.6] | 77.0 [56.1 to 105.7]
  Year 13 (N = 77;92) | 92.4 [65.9 to 129.5] | 70.1 [51.2 to 96.0]
  Year 14 (N= 75;91) | 81.8 [57.5 to 116.4] | 70.2 [51.0 to 96.8]
  Year 15 (N= 74;88) | 87.2 [61.0 to 124.5] | 69.6 [50.0 to 96.9]

4. Primary Outcome: Anti-HBs Anamnestic Response.
Description: Anamnestic response was defined as:
  Anti-HBs antibody concentrations ≥ 10 mIU/mL at one month post-challenge dose in subjects seronegative at the pre-challenge time-points.
  At least a 4-fold increase in anti-HBs antibody concentrations, at one month post-challenge dose in subjects seropositive at the pre-challenge time-points.
Time Frame: One month after the challenge dose.
Population: Analysis was performed on Total Vaccinated cohort for challenge dose that included all subjects who received the challenge dose and for whom the immunogenicity data were available.
Measure: Number; unit: Subjects
Arm/Group | Twinrix Adult Group | Twinrix Junior Group
Number analyzed (Participants) | 8 | 11
Subjects | 8 | 10

5. Primary Outcome: Number of Subjects With Anti-Hepatitis A (HAV) Antibody Concentrations Equal to or Above the Cut-Off Value.
Description: Anti-HAV antibody cut-off value assessed was >= 15 milli-International Units per milliliter (mIU/mL).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: subjects
Arm/Group | Twinrix Adult Group | Twinrix Junior Group
Number analyzed (Participants) | 78 | 92
subjects
  Year 11 (N= 78; 92) | 78 | 92
  Year 12 (N= 75; 90) | 75 | 90
  Year 13 (N= 77; 92) | 76 | 92
  Year 14 (N= 75; 91) | 75 | 91
  Year 15 (N= 74; 88) | 74 | 88

6. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs) or Hepatitis A or B Infection.
Description: SAE is any untoward medical occurrence that: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
Time Frame: Since the last long-term follow-up visit up to Year 11.
Population: Analysis was performed on Long Term (LT) Total Cohort which included all subjects who returned at the current follow-up study and who belonged to the Total cohort in the primary study.
Measure: Number; unit: subjects
Arm/Group | Twinrix Adult Group | Twinrix Junior Group
Number analyzed (Participants) | 99 | 111
subjects | 0 | 0

7. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs) or Hepatitis A or B Infection.
Description: as for outcome 6
Time Frame: Since the last long-term follow-up visit up to Year 12.
Population: as for outcome 6
Measure: Number; unit: subjects
Arm/Group | Twinrix Adult Group | Twinrix Junior Group
Number analyzed (Participants) | 101 | 109
subjects | 0 | 0

8. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs) or Hepatitis A or B Infection.
Description: as for outcome 6
Time Frame: Since the last long-term follow-up visit up to Year 13.
Population: as for outcome 6
Measure: Number; unit: subjects
Arm/Group | Twinrix Adult Group | Twinrix Junior Group
Number analyzed (Participants) | 102 | 113
subjects | 0 | 0

9. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs) or Hepatitis A or B Infection.
Description: as for outcome 6
Time Frame: Since the last long-term follow-up visit up to Year 14.
Population: as for outcome 6
Measure: Number; unit: Subjects
Arm/Group | Twinrix Adult Group | Twinrix Junior Group
Number analyzed (Participants) | 100 | 113
Subjects | 0 | 0

10. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs) or Hepatitis A or B Infection.
Description: as for outcome 6
Time Frame: Since the last long-term follow-up visit up to Year 15.
Population: as for outcome 6
Measure: Number; unit: Subjects
Arm/Group | Twinrix Adult Group | Twinrix Junior Group
Number analyzed (Participants) | 98 | 111
Subjects | 0 | 0

11. Secondary Outcome: Number of Subjects With Anti-hepatitis A (HAV) Antibody Concentrations Equal to or Above the Cut-off Value.
Description: Anti-HAV antibody cut-off value assessed was >= 15 milli-International Units per milliliter (mIU/mL).
  Note: Since none of the subjects were seronegative for anti-HAV antibody concentration at the pre-challenge time point, subjects received only the HBV vaccine as the challenge dose.
Time Frame: Before (PRE) the challenge dose
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Twinrix Adult Group | Twinrix Junior Group
Number analyzed (Participants) | 8 | 11
Subjects | 8 | 11

12. Secondary Outcome: Anti-HAV Antibody Concentrations
Description: as for outcome 1
Time Frame: Before (PRE) the challenge dose
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Twinrix Adult Group | Twinrix Junior Group
Number analyzed (Participants) | 8 | 11
mIU/mL | 270.9 [173.8 to 422.3] | 201.3 [123.1 to 329.0]

13. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Adverse Events.
Description: Solicited local symptoms assessed were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site.
Time Frame: During the 4-day (Day 0 to Day 3) follow-up period after the challenge dose
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Twinrix Adult Group | Twinrix Junior Group
Number analyzed (Participants) | 8 | 11
Subjects
  Any Pain | 5 | 4
  Grade 3 Pain | 0 | 0
  Any Redness | 1 | 2
  Grade 3 Redness | 0 | 0
  Any Swelling | 0 | 0
  Grade 3 Swelling | 0 | 0

14. Secondary Outcome: Number of Subjects With Anti-hepatitis B Surface Antigen (HBs) Antibody Concentrations Equal to or Above the Cut-off Values
Description: Anti-HBs antibody cut-off values assessed were >= 6.2 mIU/mL and >= 10 mIU/mL
Time Frame: Before (PRE) and one month after (POST) the challenge dose
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Twinrix Adult Group | Twinrix Junior Group
Number analyzed (Participants) | 8 | 11
Subjects
  PRE [6.2 mIU/mL] (N = 8;11) | 0 | 2
  POST [6.2 mIU/mL] (N = 8;11) | 8 | 11
  PRE [10 mIU/mL] (N = 8;11) | 0 | 1
  POST [10 mIU/mL] (N = 8;11) | 8 | 10

15. Secondary Outcome: Anti-HBs Antibody Concentrations
Description: Antibody concentrations are expressed as Geometric Mean concentrations (GMCs) in mIU/mL. The analysis was performed on anti-HBs seropositive subjects. Seropositive subjects are subjects with anti-HBs antibody concentrations >= 6.2 mIU/mL.
Time Frame: Before (PRE) and one month after (POST) the challenge dose
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Twinrix Adult Group | Twinrix Junior Group
Number analyzed (Participants) | 8 | 11
mIU/mL
  PRE (N= 8;11) | 3.1 [3.1 to 3.1] | 4.1 [2.5 to 6.9]
  POST (N= 8;11) | 3022.8 [407.8 to 22405.5] | 1433.1 [324.5 to 6328.9]

16. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms.
Description: Solicited general symptoms assessed were fatigue, gastrointestinal symptoms, headache and fever (axillary temperature). Gastrointestinal symptoms included nausea, vomiting, diarrhoea and/or abdominal pain. Any = occurrence of any general symptom regardless of intensity grade or relationship to vaccination. Grade 3 symptoms = symptoms that prevented normal activity. Grade 3 fever = axillary temperature > 39.5°C. Related = general symptoms which were assessed by the investigator as causally related to vaccination.
Time Frame: During the 4-day (Day 0 to Day 3) follow-up period after the challenge dose.
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Twinrix Adult Group | Twinrix Junior Group
Number analyzed (Participants) | 8 | 11
Subjects
  Any Fatigue | 3 | 3
  Grade 3 Fatigue | 0 | 0
  Related Fatigue | 3 | 3
  Any Gastrointestinal symptoms | 1 | 1
  Grade 3 Gastrointestinal symptoms | 0 | 0
  Related Gastrointestinal symptoms | 1 | 1
  Any Headache | 1 | 2
  Grade 3 Headache | 0 | 0
  Related Headache | 1 | 2
  Any Temperature | 0 | 0
  Grade 3 Temperature | 0 | 0
  Related Temperature | 0 | 0

17. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited Symptoms.
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any was defined as an adverse event (AE) reported in addition to those solicited during the clinical study. Any solicited symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited adverse event. Grade 3 = AE that prevented normal activity. Related = AE assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 31-day (Day 0 to 30) follow-up period after the challenge dose.
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Twinrix Adult Group | Twinrix Junior Group
Number analyzed (Participants) | 8 | 11
Subjects
  Any AE(s) | 4 | 0
  Grade 3 AE(s) | 0 | 0
  Related AE(s) | 0 | 0

18. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs).
Description: Serious adverse events (SAEs) assessed included medical occurrences that resulted in death, were life threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: One month after the administration of the challenge dose (Month 0 to Month 1)
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Twinrix Adult Group | Twinrix Junior Group
Number analyzed (Participants) | 8 | 11
Subjects | 1 | 0

ADVERSE EVENTS:
Time Frame: SAEs: one month post challenge dose and up to Year 15 of the long-term follow-up, solicted symptoms: during the 4-day (Days 0-3) post challenge dose and unsolicited AEs: within the 31-day (Days 0-30) post challenge dose.
Description: No Serious Adverse Events (SAEs) related to primary vaccination or to lack of vaccine efficacy were reported during this long-term follow-up study up to Year 15. Other (non-serious) adverse events were not assessed for the long-term follow-up phase (up to Year 15) as per protocol.
Arm/Group | Twinrix Adult Group | Twinrix Junior Group
Serious Adverse Events (participants affected / at risk) | 1/102 | 0/113
Other Adverse Events (participants affected / at risk) | 8/8 | 7/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Twinrix Adult Group (N=102) | Twinrix Junior Group (N=113)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 — One month after the administration of the challenge dose (Month 0 to Month 1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Twinrix Adult Group (N=8) | Twinrix Junior Group (N=11)
Pain (General disorders) | 5 | 4
Redness (General disorders) | 1 | 2
Fatigue (General disorders) | 3 | 3
Gastrointestinal symptoms (Gastrointestinal disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 3 | 0

LIMITATIONS AND CAVEATS:
A decrease in the specificity of the anti-HB ELISA assay had been observed in some studies for low levels of antibody (10-100 mIU/mL).The table shows updated results following complete retesting and reanalysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.